CLINICAL TRIAL: NCT06101043
Title: Study on the PECS II Block With Postoperative Pain in Patients Undergoing Single Port Robot-assisted Transaxillary Thyroidectomy: Double-blinded Randomized Controlled Trial
Brief Title: PECS II Block and Single Port Robot-assisted Transaxillary Thyroidectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Min Suk Chae (Other)
Responsible Party: Sponsor-Investigator, Min Suk Chae, Assistant professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KC22EISI0542
Record Dates: First submitted 2023-10-19; First posted 2023-10-25 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PECS II block group (Experimental)
  Interventions: Procedure: Pectoral nerve block
- No PECS II block group (No Intervention)

INTERVENTIONS:
Procedure: Pectoral nerve block — An ultrasound probe was placed obliquely over the second and third ribs below the lateral one-third of the clavicle. After identification of the anatomical structures, the needle was advanced along a superior-medial-to-inferior-lateral passage to the tissue plane between the pectoralis minor and serratus anterior muscles, and 20 mL ropivacaine (0.375% w/v) was injected at the level of the third rib. The anesthetic spread around the axilla, and the needle was withdrawn to the point in the plane between the pectoralis major and minor muscles. A second injection of 20 mL ropivacaine (0.375% w/v) was then delivered (PECS II).
  Arms: PECS II block group

SUMMARY:
The da Vinci robotic system was developed to improve both operative maneuverability (through multi-articulated instruments) and the surgical view (via a three-dimensional camera). Although the system has many advantages, skin incision, wide flap dissection, and pneumatic/mechanical retraction remain essential, but cause postoperative pain and slower recovery. Previous studies found that pectoralis fascial blocks were easy to establish; local anesthetics are injected between two adjacent myofascial layers under ultrasound guidance, providing the surgeon with a clear image. Analgesic efficacy has been validated during robotic thyroidectomy in our institution. The pain outcomes were comparable between the groups, but there were fewer complications in the PECS II group. The investigators investigated whether this block can reduce postoperative pain during wide flap dissection for single-port robot-assisted transaxillary thyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 to 60 years who are scheduled to undergo single-port robot thyroidectomy (lobectomy or total thyroidectomy)
* Patients with cancer stages T1 or T2 (less than 4 cm without invasion of surrounding tissue) when thyroid cancer is suspected in the preoperative examination
* Patients with nodules with a maximum length of less than 4 cm based on ultrasonography if thyroid cancer is not suspected in the preoperative examination
* Patients with a BMI greater than or equal to 18.5 and less than 30.0.

Exclusion Criteria:

* Patients requiring lateral cervical lymph node dissection
* pregnant women
* Uncontrolled diabetes
* Chronic kidney failure
* Patients with previous neck surgery
* Patients with Graves' disease
* People with chronic alcoholism
* Patients with vocal cord paralysis before surgery
* Severe obese patients with a body mass index >35 kg/m2
* Patients participating in another clinical trial within 30 days
* Patients who expect that it will be difficult for medical staff to fill out the questionnaire on their own
* Patients whose medical staff determines that participation in the study is difficult due to other underlying diseases

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-01-04 (Estimated); Primary Completion 2024-09-28 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Analgesic efficacy | the day after surgery
  Visual analog scale from 0 (minimum) to 10 (maximum)

SECONDARY OUTCOMES:
Quality of postoperative surgery course | the day after surgery
  The Korean version of QoR-15 (QoR-15K questionnaire) from 0 (minimum) to 150 (maximum)